CLINICAL TRIAL: NCT00713960
Title: CARE - Quality Development in Cardiovascular Disease in General Practice
Brief Title: CARE - Quality Improvement in Cardiovascular Secondary Prevention in Primary Care, Through Delegation of Consultations to the Nurse.
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS-CDK-DUM-2008/1
Record Dates: First submitted 2008-07-10; First posted 2008-07-14 (Estimated); Last update posted 2012-01-16 (Estimated); Status verified 2012-01

CONDITIONS: Cardiovascular Disease
Keywords: Quality development project; primary care nurses; cardiovascular disease; secondary prevention; follow-up
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Patients in secondary prevention of cardiovascular disease in primary care

SUMMARY:
Quality Improvement in Primary Care: delegation of check-ups to nurses in general practice

ELIGIBILITY:
Inclusion Criteria:

* Patients in secondary prevention of cardiopathy (ischaemic heart disease, claudication intermittence, thrombotic apoplexy cerebri, diabetes) who are not followed in an outpatient department.

Exclusion Criteria:

* Patients who suffer from diabetic nephropathy will be excluded
* According to the general practitioners appraisal, patients who suffer from severe co morbidity can be excluded as well.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 2193 (Actual)
Dates: Start 2008-04; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Cholesterol, HDL -cholesterol, LDL-Cholesterol, Blood pressure, Exercise, Waist-circumference, BMI, Smoking status, fasting plasma-glucose, medication taken | As needed, min. baseline and after 6 months

SECONDARY OUTCOMES:
Number of visits pr. patients, drop-out | Annually

CONTACTS AND LOCATIONS:
Overall Officials: Henrik Ommen, MD, Study Chair — Lægerne i Løgumkloster I/S, Denmark; Dorte Knudsen, Study Chair — Lægerne Sønderåparken, Denmark
Locations (66):
- Denmark (66):
  - Research Site, Albertslund
  - Research Site, Arhus C
  - Research site, Assens
  - Research Site, Billund
  - Research Site, Brabrand
  - Research Site, Elsinore
  - Research Site, Erslev
  - Research Site, Esbjerg
  - Research Site, Faaborg
  - Research Site, Gentofte Municipality
  - Research Site, Give
  - Research Site, Greve
  - Research Site, Hadsund
  - Research Site, Hedehusene
  - Research Site, Hillerød
  - Research Site, Hinnerup
  - Research Site, Hjallerup
  - Research Site, Hjørring
  - Research Site, Hobro
  - Research Site, Holaek
  - Research Site, Holstebro
  - Research Site, Hornsyld
  - Research Site, Horsens
  - Research Site, Hørning
  - Research Site, Karup
  - Research Site, Kbh. O
  - Research Site, Kerteminde
  - Research Site, Kjellerup
  - Research Site, Klarup
  - Research site, Kobenhavn V
  - Research Site, Kolding
  - Research Site, Kolding C
  - Research Site, Kongens Lyngby
  - Research Site, København Ø
  - Research Site, Køge
  - Research Site, Lemvig
  - Research Site, Lystrup
  - Research Site, Maribo
  - Research Site, Nivå
  - Research Site, Næstved
  - Research Site, Odense C
  - Research Site, Pandrup
  - Research Site, Randers
  - Research Site, Ringsted
  - Research Site, Roskilde
  - Research Site, Rungsted Kyst
  - Research Site, Rødding
  - Research Site, Silkeborg
  - Research Site, Skælskør
  - Research Site, Solrød Strand
  - Research Site, Stege
  - Research Site, Struer Municipality
  - Research Site, Svendborg
  - Research Site, Svinninge
  - Research Site, Sønder Felding
  - Research Site, Sønderborg
  - Research Site, Thisted
  - Research Site, Tune
  - Research Site, Vamdrup
  - Research Site, Varde
  - Research Site, Vejen Municipality
  - Research Site, Vejle
  - Research Site, Vestervig
  - Research Site, Viborg
  - Research Site, Viby J
  - Research Site, Vivild